CLINICAL TRIAL: NCT06665334
Title: Objective to Explore the Effect of Huaier Granule on the Negative Conversion Rate of Patients Whose Carcinoembryonic Antigen (CEA) Level Increases Again After Radical Resection of Colorectal Cancer
Brief Title: To Explore the Effect of Huaier Granule on the Negative Conversion Rate After the CEA Level Increases Again After Colorectal Cancer Surgery
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ye Xu, professor, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HE-202203
Record Dates: First submitted 2024-10-29; First posted 2024-10-30 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Colorectal Cancer
Keywords: Huaier Granule; Colorectal Cancer; CEA Level; Negative Conversion Rate
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Huaier Granule (Experimental): Oral administration of Huaier granule, 10g (1 bag) each time, 3 times a day, is recommended for at least 6 months until there is imaging progression of the disease, the end of the study, intolerable toxicity, withdrawal or death from the study for any reason, or the researcher determines that there is no longer benefit, whichever occurs first.
  Interventions: Drug: Huaier granule
- Routine clinical treatment (No Intervention): During routine clinical follow-up, patients who underwent R0 resection were found to have abnormally elevated levels of CEA, and therefore no intervention was generally given. If there is imaging progress, intolerable toxicity, or withdrawal from the study for any reason during the research period (whichever occurs first), routine clinical treatment will be administered.

INTERVENTIONS:
Drug: Huaier granule — Oral administration, 10g per dose (1 bag), 3 times a day, recommended for at least 6 months.
  Other Names: Z20000109#NMPA Approval Number#
  Arms: Huaier Granule

SUMMARY:
This study is a prospective, observational and exploratory study to explore the effect of Huaier Granule on the negative conversion rate of patients with increased CEA levels after colorectal cancer surgery.

DETAILED DESCRIPTION:
This study is a prospective, single center, observational study, expected to include patients who visited the selected research center from December 2022 to December 2024 and were pathologically diagnosed with stage I-III colorectal cancer and underwent R0 radical resection surgery. During routine clinical follow-up within one year after radical surgery, if serum CEA>5.2ng/ml occurs, patients may choose whether to use Huaier granules to prevent recurrence and metastasis according to their wishes. Patients who agree to use Huaier granules will enter the observation group; Patients who do not agree to use it will enter the control group. After the subjects are enrolled, they will be visited every 1 month ± 7 days in the first year, and every 3 months ± 14 days starting from the second year according to clinical routine diagnosis and treatment, until imaging examination determines disease progression, the end of the study, intolerable toxicity, withdrawal from the study for any reason or death, or the researcher determines no longer benefiting, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old, gender not limited
* Diagnosed with colorectal cancer through histopathology, pTNM stage I-III
* Previously underwent radical resection for colorectal cancer, with a postoperative evaluation of R0
* Imaging did not detect recurrence or distant metastasis
* Serum CEA>5.2ng/ml within 1 year after surgery (found during routine clinical follow-up)
* Clear consciousness, language expression or reading ability, able to communicate normally, and cooperate to complete the questionnaire evaluation
* Voluntary participation in this study, good compliance, and signing of informed consent form.

Exclusion Criteria:

* Known to be allergic to the components of Huaier Granule, or to avoid or use Huaier Granule with caution (observation group)
* Cannot take medicine orally
* Have received anti-tumor traditional Chinese patent medicines and simple preparations treatment within 1 month before enrollment (subject to the instructions)
* Combining medical history of other malignant tumors
* Diabetes with serious heart, cerebrovascular and lung diseases, severe hypertension and poor blood sugar control
* Suffering from intestinal diverticulitis, rectal polyps, colitis, pancreatitis, cirrhosis, hepatitis, etc
* Currently participating in clinical trials of other drugs
* Pregnant or lactating women or those planning to conceive
* Refusing to cooperate with follow-up visits
* Other reasons led the investigators to believe that it was not suitable to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Rate of CEA conversion to negative | start of treatment until 2-year follow-up
  The proportion of patients whose CEA levels returned to normal at each visit to the total number of patients at that follow-up.

SECONDARY OUTCOMES:
1 or 2-year disease-free survival rate (DFS) | start of treatment until 2-year follow-up
  The proportion of surviving patients who did not experience imaging recurrence, distant metastasis, or death within 1 or 2 years after enrollment.
Quality of Life Score | baseline period and start of treatment until 2-year follow-up
  Evaluation using the EORTC QLQ-C30 (Chinese version) core quality of life scale developed by the European Organization for Cancer Research and Treatment.

OTHER OUTCOMES:
The changes (rate values) of tumor markers (including but not limited to CA199, CA24-2, CA72-4, and CA50) compared to baseline | start of treatment until 2-year follow-up
  The differences in tumor marker levels between treatment and baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Ye Xu, PhD, Principal Investigator — Fudan University